CLINICAL TRIAL: NCT04778956
Title: Toripalimab Plus Surgery vs Surgery Alone for Resectable Recurrent Nasopharyngeal Carcinoma: a Prospecitve, Parallel, Multicenter, Phase III, Randomized Clinical Trial
Brief Title: Toripalimab Plus Surgery vs Surgery Alone for Resectable Recurrent Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Nanfang Hospital, Southern Medical University (Other); First People's Hospital of Foshan (Other); Zhongshan People's Hospital, Guangdong, China (Other); Tenth Affiliated Hospital, Sun Yat-sen University (Unknown)
Responsible Party: Principal Investigator, Ming-Yuan Chen, Professor, Chief Doctor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-CMY-2020-2302
Record Dates: First submitted 2021-02-25; First posted 2021-03-03 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Nasopharyngeal Carcinoma; PD-1; Surgery
Keywords: Nasopharyngeal carcinoma; Recurrent; Salvage surgery; Anti-programmed death-1 antibody; Disease free survival
MeSH Terms: conditions — Nasopharyngeal Carcinoma; Recurrence | interventions — toripalimab; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Toripalimab plus salvage surgery (Experimental): 1. Toripalimab: Toripalimab treatment before and after salvage surgery.
  2. Salvage surgery: endoscopic nasopharyngectomy for recurrent nasopharyngeal tumor, and selective neck dissection for recurrent regional lymph node.
  Interventions: Drug: Toripalimab; Procedure: salvage surgery
- Salvage surgery alone (Active Comparator): 1. Salvage surgery: endoscopic nasopharyngectomy for recurrent nasopharyngeal tumor, and selective neck dissection for recurrent regional lymph node.
  Interventions: Procedure: salvage surgery

INTERVENTIONS:
Drug: Toripalimab — Toripalimab: 240 mg, intravenous injection over 60 minutes (Q3W); Toripalimab should be completed for 2 cycles at 1-2 weeks before surgery, and continually applied since 1-2 weeks after surgery until confirmed disease progression, death, unacceptable toxicity, withdrawal of consent, investigator decision, or 1 year.
  Other Names: PD-1 antibody
  Arms: Toripalimab plus salvage surgery
Procedure: salvage surgery — Endoscopic nasopharyngectomy is used for recurrent nasopharyngeal tumor and selective neck dissection for recurrent regional lymph node.

SUMMARY:
Through multicenter, open-label, randomised clinical trials, we intend to demonstrate that PD-1 treatment added to salvage surgery could further decrease the rate of disease progression and improve the survival outcome of patients with resectable locally recurrent nasopharyngeal carcinoma compared with those treated with salvage surgery alone.

DETAILED DESCRIPTION:
Through multicenter, open-label, randomised clinical trials, patients with resectable locally recurrent nasopharyngeal carcinoma are randomized into salvage surgery plus PD-1 treatment group and salvage surgery alone group. The efficacy and safety of patients between these two groups are compared.

ELIGIBILITY:
Inclusion Criteria:

1. The recurrence time is more than 6 months from the end of radiotherapy.
2. Histologically confirmed recurrent nasopharyngeal carcinoma.
3. Resectable nasopharyngeal diseases: recurrent T1 (the tumor is confined in nasopharynx, oropharynx and/or nasal cavity without parapharyngeal involvement); recurrent T2 (the tumor is confined in the superficial parapharyngeal spacer and is more than 0.5cm far from the internal carotid artery) and recurrent T3 (the tumor is confined in the base wall of the sphenoid sinus and is more than 0.5cm far from the internal carotid artery and cavernous sinus). (according to the 8th edition of American Joint Committee on Cancer (AJCC) staging system for nasopharyngeal carcinoma)
4. Resectable recurrent regional lymph node diseases (recurrent N1-3) without prevertebral fascia, cervical vertebrae, or common/internal carotid artery involvement. (according to the 8th edition of AJCC staging system)
5. Given written informed consent.

Exclusion Criteria:

1. Karnofsky Performance Status (KPS) ≤70.
2. Has severe medical disorder, important organ dysfunction, and/or a substantial history of mental illness.
3. Has known subjects with other malignant tumors.
4. Has participated in other drug trials within 3 months of planned start of study treatment.
5. Received a systematic or local glucocorticoid therapy within 4 weeks of planned start of study treatment.
6. Suffered from diseases need long-term treatment with immunosuppressive drugs, or required systematic or local glucocorticoid therapy with immunosuppressive doses.
7. Prior therapy with a PD-1, anti-PD-Ligand 1 (PD-L1) or cytotoxic T lymphocyte-associated antigen 4 (CTLA-4) agent.
8. Has active autoimmune disease (e.g., uveitis, enteritis, hepatitis, hypophysitis, nephritis, vasculitis, hyperthyroidism, and asthma requiring bronchodilator therapy). Patients with skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia) will be allowed to enroll.
9. Has a known history of human immunodeficiency virus (HIV), has hepatitis B surface antigen (HBsAg) positive with hepatitis B virus (HBV) DNA copy number of ≥1000cps/ml or hepatitis C virus (HCV) antibody positive.
10. Has received a live vaccine within 4 weeks of planned start of study treatment.
11. Pregnancy or breast feeding.
12. Cannot complete regular follow-up.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Estimated)
Dates: Start 2021-03-03 (Actual); Primary Completion 2025-03-03 (Estimated); Study Completion 2033-03-03 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 2 years
  Defined as the time interval from randomization to disease progression or death due to any cause, whichever come first.

SECONDARY OUTCOMES:
Objective Response Rate | 3-5 weeks
  Defined as the proportion of patients with radiologically confirmed complete or partial response according to RECIST 1.1.
Major Pathological Response Rate | 4-6 weeks
  Defined as the proportion of patients with no more than 10% viable tumor cells which is identified on routine hematoxylin and eosin staining within the recurrent nasopharyngeal tumor and/or regional lymph node after neoadjuvant PD-1 treatment.
Overall Survival | 2 years
  Defined as the time interval from randomization to death due to any cause.
Distant Metastasis-Free Survival | 2 years
  Defined as the time interval from randomisation to the date of first distant metastases.
Locoregional Relapse-Free Survival | 2 years
  Defined as the time from randomisation to the date of first locoregional relapse.
Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) | up to 2 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire (QLQ)-C30 (V3.0) before treatment, during treatment, after treatment.
Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) | up to 2 years
  Score of survival quality according to the EORTC Quality of Life Questionnaire Head and Neck (The QLQ-H&N35) before treatment, during treatment, after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Yuan Chen, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (7):
- China (7):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First People's Hospital of Foshan, Guangzhou, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - The Tenth Affiliated Hospital, Sun Yat-Sen University, Nanchang, Jiangxi